CLINICAL TRIAL: NCT06817720
Title: Phase II Study Assessing the Efficacy and Toxicity of Olverembatinib Monotherapy in Patients With Newly Diagnosed Chronic Myeloid Leukemia in Chronic Phase
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Ascentage Pharma Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1637; NCI-2025-00934 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — olverembatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment with Olveremebatinib (Experimental): Patients will receive single agent olverembatinib at a dose of 30 mg orally every other day (QOD)
  Interventions: Drug: olverembatinib

INTERVENTIONS:
Drug: olverembatinib — GIven by PO

SUMMARY:
To learn if olverembatinib can help to control newly diagnosed CML in the chronic phase.

DETAILED DESCRIPTION:
Primary Objectives

* To assess the rate of MMR by 12 months. Secondary Objectives
* To assess the rate of CCyR by 12 months.
* To estimate the proportion of participants with 4.5-log reduction of BCR::ABL1 transcripts (MR4.5) at 6, 12, 18, 24, and 36 months of therapy.
* To estimate the rate of sustained deep molecular response.
* To estimate event-free survival and overall survival.
* To assess the toxicity of olverembatinib monotherapy.
* To assess health-related quality of life (HRQOL) of the participants.

ELIGIBILITY:
Eligibility Criteria:

* Adult participants age ≥18 years.
* Participants must have a diagnosis of Ph-positive or BCR::ABL1 positive CML in early chronic phase.
* Participants who received prior hydroxyurea, 1 to 2 doses of cytarabine, and/or an FDA approved TKI for ≤ 30 days are eligible.
* Participants with additional chromosomal abnormalities at diagnosis (early disease) and no other criteria for accelerated phase will be eligible for this study.
* ECOG performance status ≤ 2.
* Participants must have adequate end organ function, defined as the following: total bilirubin ≤1.5x ULN (unless secondary to Gilbert's disease, in which case should be ≤ 2.5x ULN), SGPT or SGOT ≤ 3x ULN, creatinine clearance ≥ 30mL/min calculated using modified Cockcroft-Gault.
* Ability to understand and the willingness to sign a written informed consent document.
* The effects of olverembatinib on the developing human fetus are unknown. For this reason,women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and 4 months after completion of olverembatinib administration. This includes all female participants, between the onset of menses (as early as 8 years of age) and 55 years unless the participants presents with an applicable exclusionary factor which may be one of the following:

  * Postmenopausal (no menses in greater than or equal to 12 consecutive months).
  * History of hysterectomy or bilateral salpingo-oophorectomy.
  * Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
  * History of bilateral tubal ligation or another surgical sterilization procedure.
* Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Participant post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

  * Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of olverembatinib administration.
  * For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
  * Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured.

For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.

* Participants with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression.
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants should be class 2 or better.

Exclusion Criteria:

* Participants who have received more than 30 days of prior FDA approved TKI or more than 2 doses of cytarabine.
* Had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study.
* Participants who have not recovered from adverse events due to prior anti-cancer therapy with the exception of alopecia.
* Participants who are receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to olverembatinib or other agents used in study.
* NYHA cardiac class 3-4 heart disease
* Cardiac Symptoms: Participants meeting the following criteria are not eligible unless cleared by cardiologist

  * Uncontrolled angina within 3 months
  * Diagnosed or suspected congenital long QT syndrome
  * Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes).
  * Prolonged QTc interval on pre-entry electrocardiogram (> 460 msec)
* History of significant bleeding disorder unrelated to cancer, including unless cleared by hematologist or hemato-oncologist:

  * Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease)
  * Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies)

    * Participants with active, uncontrolled psychiatric disorders including psychosis, major depression, and bipolar disorders.
    * Participants with cognitive impairment or psychiatric illness/social situations that would limit compliance with study requirements.
    * Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
    * Evidence of other clinically significant uncontrolled condition(s) including, but not limited to:
  * Uncontrolled and/or active systemic infection (viral, bacterial or fungal)
  * Chronic hepatitis B virus (HBV) or hepatitis C (HCV) requiring treatment and having detectable virus load. Note: subjects with serologic evidence of prior vaccination to HBV (i.e. hepatitis B surface antigen negative, anti-HBs antibody positive and antihepatitis B core antibody negative) or positive anti-HBc antibody from intravenous immunoglobulins may participate.

    * Pregnant women are excluded from this study because olverembatinib is a BCR::ABL1 TKI with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with olverembatinib, breastfeeding should be discontinued if the mother is treated with olverembatinib. These potential risks may also apply to other agents used in this study.
    * Participants in late chronic phase (i.e., time from diagnosis to treatment > 12 months), accelerated (except as noted in inclusion criteria 4.1) or blast phase are excluded. The definitions of CML phases are as follows:
  * Early chronic phase: time from diagnosis to therapy ≤ 12 months.
  * Late chronic phase: time from diagnosis to therapy > 12 months.
  * Blastic phase: presence of 30% blasts or more in the peripheral blood or bone marrow.
  * Accelerated phase CML: presence of any of the following features:

    i. Peripheral or marrow blasts 15% or more. ii. Peripheral or marrow basophils 20% or more. iii. Thrombocytopenia < 100 x 109/L unrelated to therapy. iv. Documented extramedullary blastic disease outside liver or spleen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2027-03-07 (Estimated); Study Completion 2027-03-07 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Fadi Haddad, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org